CLINICAL TRIAL: NCT03735004
Title: The Effects of Transcranial Electrostimulation (TES) on Postoperative Pain and Functional Patient Outcomes After Surgery for Obstructive Sleep Apnea Syndrome
Brief Title: Transcranial Electrostimulation and Obstructive Sleep Apnea Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vladimir Nekhendzy, Clinical Professor of Anesthesiology and Otolaryngology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 29984
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Transcranial Electrical Stimulation
Keywords: electrical stimulation; electric anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- TES 60 Hz DC:AC (Experimental): Transcranial electrostimulation (TES) with combined direct (DC) and alternating (AC, 60 Hz) current
  Interventions: Device: Transcranial electrostimulation (TES)
- TES 100 Hz DC:AC (Active Comparator): Transcranial electrostimulation (TES) with combined direct (DC) and alternating (AC, 100 Hz) current
  Interventions: Device: Transcranial electrostimulation (TES)
- TES with DC current (Sham Comparator): Transcranial electrostimulation (TES) with direct current (DC) only
  Interventions: Device: Transcranial electrostimulation (TES)

INTERVENTIONS:
Device: Transcranial electrostimulation (TES) — Transcranial electrostimulation (TES) with combined direct (DC) and alternating (AC) current, or TES with DC only will be administered through the skin electrodes positioned on the patient's head

SUMMARY:
Postoperative pain after major surgery for obstructive sleep apnea (OSA), such as palatopharyngoplasty (PPP) and maxillomandibular advancement (MMA) is moderate-to-severe, and may persist for weeks. Control of this pain may be difficult, because OSA patients are very sensitive to traditional opioid pain medications, and their side effects. Poorly controlled pain slows down patients' recovery after surgery, including a return to normal daily activities and work, and may also delay wound healing.

This study will investigate whether pain relief and recovery after surgery may be improved with the application of a weak electrical current to the skin of the patient's head (transcranial electrostimulation, TES). The TES works by blocking pain in the central nervous system through multiple mechanisms, which result in non-pharmacological pain relief, without drug-associated side effects.

DETAILED DESCRIPTION:
The incidence and severity of postoperative pain in patients undergoing major airway surgery for OSA, such as palatopharyngoplasty (PPP) and maxillomandibular advancement (MMA) is high, and may persist for days, significantly contributing to patient's morbidity. High doses of intravenous and oral opioids are frequently required to achieve adequate pain relief. Yet, the increased sensitivity of OSA patients to opioid analgesics, and associated high risk of postoperative respiratory depression and upper airway obstruction limit the traditional therapeutic options, frequently making pain control after PPP and MMA surgery suboptimal.

The effect of significant postoperative pain on surgical outcomes is multifold. Poorly controlled post-surgical pain increases patient morbidity, impairs wound healing, and negatively affects patient recovery and functional outcomes, such as ambulation, a resumption of a normal oral intake, a return to normal daily activities, a return to work, and others. Side effects of opioid medications, such as urinary retention, constipation, nausea, vomiting, dizziness, and itching may further adversely affect recovery and cause patient dissatisfaction with the surgical procedure.

The development of the new, effective analgesic modalities, is therefore highly desirable for OSA surgical patients, and particularly those undergoing PPP and MMA surgeries. Transcranial electrostimulation (TES) is a non-invasive brain stimulation technique that employs administration of a weak electrical current (≤ 5 mA) through the electrodes positioned on the skin of the patient's head. TES is a safe procedure, with a low risk of associated, minor side effects It is widely believed that TES with combined direct (DC) and alternating (AC) current (TES DC:AC) triggers the release of endogenous opioids and other central neurotransmitters (e.g. norepinephrine) that interrupt nociceptive processing. The investigator's previous studies have demonstrated that TES DC:AC produces quickly evolving, effective non-pharmacological analgesia, without associated respiratory depression or other opioid-induced side effects. If analgesic effect of TES can be demonstrated in this study, the TES may become an attractive adjunct for postoperative analgesic treatment for OSA patients, allowing for improved quality of analgesia and enhanced recovery.

Moreover, demonstrating TES analgesic effect may facilitate its widespread use as a non-pharmacological analgesic adjunct postoperatively, especially in elderly patients, who have a high incidence of associated OSA and sensitivity to systemic opioids. The incidence of OSA in general surgical population reaches over 20%.

ELIGIBILITY:
Inclusion Criteria: Patients with moderate-to-severe OSA, presenting for PPP and MMA surgeries. All patients will be American Society of Anesthesiology (ASA) physical status II-III. The subjects should understand informed consent and study instructions.

Exclusion Criteria:

1. Patients with a known or suspected genetic susceptibility to malignant hyperthermia, or known sensitivity to Sevoflurane, an inhaled anesthetic agent.
2. Pregnant patients.
3. Patients who are unable to understand the questionnaires or the visual analogue scale (VAS) pain scores, or to keep home diaries.
4. Patients with clinically-significant psychological disorders, psychiatric illness or treatment.
5. Alcohol and drug-abusing patients.
6. Patients with the history of seizures.
7. Patients with the documented or suspected organic brain or psychiatric disease, in particular with the history of hallucinations and delusions.
8. Patients with history of significant eye disease, or head or eye injury, which led to alteration of the cranial anatomy or metallic intracranial implants.
9. Patients with the history of significant surgery of the head and/or eye.
10. Patients with skin lesions and/or defects over the areas where TES electrodes will be applied.
11. Patients with implanted medical devices, including cardiac pacemakers.
12. Patients who participate in other research protocols that may interfere with the study outcomes and objectives.
13. Other patients that may be excluded by the investigator, based on medical history and physical examination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Opioid requirements during first postoperative TES session | Recorded during a 20 min TES session administered for first moderate-to-severe postoperative pain in the recovery room
  IV morphine milligram equivalents
Pain scores during first postoperative TES session | Recorded during a 20 min TES session administered for first moderate-to-severe postoperative pain in the recovery room
  VAS pain scores (Pain measured using 11-point visual analog scale 0-10, 0 no pain, 10 worst pain imaginable).
Postoperative opioid consumption during recovery room stay | Through the recovery room stay, on average 2.5 hours
  IV morphine milligram equivalents
Postoperative pain scores during recovery room stay | Through the recovery room stay, on average 2.5 hours
  VAS pain scores

SECONDARY OUTCOMES:
Postoperative opioid consumption during hospital stay | From "floor ready" until hospital discharge, on average 2 days
  PO morphine milligram equivalents
Post-discharge postoperative opioid consumption | From hospital discharge to up to 4 weeks postoperatively
  PO morphine milligram equivalents
Time to start of soft diet | Day of surgery to starting a soft diet (up to 7 days)
Time to return to daily activities | Day of surgery to return to daily activities (up to 10 days)
Time to return to work | From the day of surgery to return to work (up to 21 days)
Change from baseline in QoR15 score (Quality of Recovery 15-question score) | Baseline (before surgery) to postoperative week 4.
  Validated multidimensional questionnaire assessing recovery profile. Each scale is scored from 0-10, overall score from 0 to 150. The higher scores indicate better recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Nekhendzy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Univeristy Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No